CLINICAL TRIAL: NCT03626077
Title: Augmented Biofeedback Training Combined With Physical Therapy Program Improves Visual-motor Integration, Visual Perception and Motor Coordination in Children With Spastic Hemiplegic Cerebral Palsy: a Randomized Control Trial
Brief Title: Biofeedback Training and Physical Therapy Program Improves Visual-motor Integration in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Princess Nourah Bint Abdulrahman University (Other)
Responsible Party: Principal Investigator, Reem M Alwhaibi, associate professor, Princess Nourah Bint Abdulrahman University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 205-S-37
Record Dates: First submitted 2018-08-04; First posted 2018-08-10 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Hemiplegic Cerebral Palsy
Keywords: Biofeedback; Visual-Motor Integration; Visual Perception

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group A (Active Comparator): Group (A) physical therapy program for 60 minutes per session, three times a week for three consecutive months
  Interventions: Other: physical therapy program
- group B (Active Comparator): Group (B) E-Link Upper Limb Exerciser (augmented biofeedback training)for 60 minutes per session, three times a week for three consecutive months
  Interventions: Device: E-Link Upper Limb Exerciser
- group C (Experimental): group (C) physical therapy program and E-Link Upper Limb Exerciser
  Interventions: Combination Product: physical therapy program and E-Link Upper Limb Exerciser

INTERVENTIONS:
Other: physical therapy program — this group received specially designed physical therapy program to facilitate eye-hand coordination and fine motor to improve VMI, VP and MC, which included: unbutton buttons, and button in all again; put the pellets in the bottle as fast as he/she can; place the shapes on its form board; build steps, wall, pyramid and a tower from cubes; cut out a line, square, triangle, and rectangular shapes on a paper by scissor; string squared cubes and lace the holes of strip.Children were trained for 60 minutes per session, three times a week for three consecutive months.
  Arms: group A
Device: E-Link Upper Limb Exerciser — The exercises in the E-Link Upper Limb Exerciser System are in the form of simple and exciting games such as soccer, hitting walls, space shooting, driving, arnd throwing balls into a bucket.Children were trained for 60 minutes per session, three times a week for three consecutive months.
  Arms: group B
Combination Product: physical therapy program and E-Link Upper Limb Exerciser — physical therapy program and E-Link Upper Limb Exerciser. Children were trained for 60 minutes per session, three times a week for three months.
  Arms: group C

SUMMARY:
The aim of this study was to investigate potential benefits of adding augmented biofeedback training to standard therapy in improving visual motor integration (VMI) visual perception (VP) and motor coordination (MC) in children with hemiplegic cerebral palsy .Participants were divided randomly into three equal groups. Group (A) received specially designed program of physical therapy intervention strategies to facilitate visual motor integration and visual perception over a period of three months. Group (B) received augmented biofeedback training only, and group (C) received augmented biofeedback training and same physical therapy program as group (A).

DETAILED DESCRIPTION:
Children were assigned randomly into three groups of equal number (A, B and C). Children were selected randomly by collecting all names of children that matched the inclusion criteria of the study then upload the names and gender using an electronic program (SPSS) which divided the sample into three equal groups (A), (B) & (C).

Group A: this group included fifteen children with spastic hemiplegic CP. Children of this group received specially designed program of physical therapy exercises to facilitate eye-hand coordination and fine motor to improve VMI, VP and MC, which included: unbutton buttons, and button in all again; put the pellets in the bottle as fast as he/she can; place the shapes on its form board; build steps, wall, pyramid and a tower from cubes; cut out a line, square, triangle, and rectangular shapes on a paper by scissor; string squared cubes and lace the holes of strip. The tools used in training program were: button strip, lacing strip and its lace, mottle with screw- on cap, markers with different colors, beads and its lacing, square cubes, pellets, papers, blunt scissors, colored cubes, different types of form board and its shapes. Adjusted chair and table were used to accommodate differences in children's body built. Children were trained for 60 minutes per session, three times a week for three consecutive months.

Group B: this group included fifteen children with spastic hemiplegic CP. Children of this group received training using the E-Link Upper Limb Exerciser for 60 minutes per session, three times a week for three consecutive months.

Group C: this group included fifteen children with spastic hemiplegic CP. Children of this group received the same physical therapy program as conducted for group A, and training with E-Link Upper Limb Exerciser as conducted for group B. The training was for 60 minutes per session, three times a week for three consecutive months.

The participated children were assessed by Beery-Buktenica Developmental Test before and after the three months of the treatment program. The average time required for evaluating each child was 40 min. The assessment and training methods were applied according to the instructions provided in the test and equipment manuals, no modifications were necessary.

ELIGIBILITY:
Inclusion Criteria:

* grade of spasticity between 1 to 1+ according to Modified ashworth Scale, the ability to handle objects independently was between level (I) and (II) according to Manual Ability Classification System (MACS), no history of epilepsy; no botulinum toxin A treatment for the upper extremities in the previous 6 months, and able to understand and follow verbal commands and instructions

Exclusion Criteria:

* presence of visual or auditory impairments, significant tightness or fixed deformities in the upper limbs, severe spasticity, autism, or severe cognitive impairment

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2017-09-03 (Actual); Primary Completion 2018-03-29 (Actual); Study Completion 2018-03-29 (Actual)

PRIMARY OUTCOMES:
Beery-Buktenica Developmental Test of Visual-Motor Integration (6th edition) "change" is being assessed | 10-15 minutes total, it is taken at baseline and after 3 months of treatment
  it evaluate the subject's ability to integrate visual and motor skills, through copying

SECONDARY OUTCOMES:
Beery-Buktenica Developmental Test- Visual Perception test. "change" is being assessed | 5 minutes, it is taken at baseline and after 3 months of treatment
  it evaluates subject visual perception (VP) and motor coordination matching shapes to stimulus form
Beery-Buktenica Developmental Test-Motor Coordination test. "change" is being assessed | 5 minutes, it is taken at baseline and after 3 months of treatment
  it evaluates subject motor coordination through tracing within a confined space

CONTACTS AND LOCATIONS:
Overall Officials: Reem M Alwhaibi, PhD, Principal Investigator — Princess Nourah Bint Abdulrahman University
Locations (1):
- Disabled Children's Association, Riyadh, Alnakeel, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
data from participants will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 12 months after study completion
Access Criteria: data access requests will be reviewed by an external independent review panel. requestors will be required to sign a data access agreement.